CLINICAL TRIAL: NCT02265393
Title: A 6-Month, Prospective, Randomized, Multicenter, Placebo-Controlled Safety Study of OTO-104 Given at 3-Month Intervals by Intratympanic Injection in Subjects With Unilateral Meniere's Disease Followed by a 6-Month Open-Label Extension
Brief Title: A 1-Year Safety Study of OTO-104 in Subjects With Unilateral Meniere's Disease Located in United Kingdom
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 104-201403
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Meniere's Disease
MeSH Terms: conditions — Meniere Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OTO-104 (Active Comparator): 12 mg OTO-104 (dexamethasone)
  Interventions: Drug: OTO-104
- Placebo (Placebo Comparator): OTO-104 vehicle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OTO-104
  Arms: OTO-104
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a 2-part study of OTO-104 in subjects with unilateral Meniere's disease in the United Kingdom. The first part is a randomized, placebo-controlled study comparing the safety profile of 2 injections of OTO-104 or placebo spaced 3 months apart. The second part is an open-label extension where all subjects will receive an additional 2 intratympanic injections of OTO-104 spaced 3 months apart. Each subject will participate on the study for a total of 1 year.

ELIGIBILITY:
Inclusion Criteria includes, but is not limited to:

* Subject has a diagnosis of definite unilateral Meniere's disease.
* Subject agrees to maintain their current standard of care treatments for Meniere's disease while on-study.

Exclusion Criteria includes, but is not limited to:

* Subject is pregnant or lactating.
* Subject has a history of immunodeficiency disease.
* Subject has a history of previous endolymphatic sac surgery.
* Subject has a history of previous use of intratympanic gentamicin in the affected ear.
* Subject has a history of drop attacks.
* Subject has experienced an adverse reaction to intratympanic injection of steroids.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Safety | Up to 1 Year
  Otoscopy, audiometry, tympanometry, adverse events

SECONDARY OUTCOMES:
Meniere's Symptom Questionnaire | Up to 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Carl LeBel, PhD, Study Chair — Otonomy, Inc.
Locations (15):
- United Kingdom (15):
  - Heatherwood & Wexham Park Hospitals, Berkshire
  - Birmingham University Hospital, Birmingham
  - BMI The Edgbaston Hospital, Birmingham
  - Southmead Hospital Bristol, Bristol
  - Oxford University Hospitals, Bucks
  - Cambridge University Hospitals, Cambridge
  - Dorset County Hospital, Dorset
  - Gloucestershire Royal Hospital, Gloucester
  - Leicester Royal Infirmary, Leicestershire
  - Guy's Hospital and St. Thomas' Hospital, London
  - St. George Hospital, London
  - Norfolk & Norwich University Hospital, Norfolk
  - John Radcliffe Hospital, Oxford
  - Sheffield Teaching Hospitals & Sheffield Children's Hospital, Sheffield
  - University Hospital of North Staffordshire, Stoke-on-Trent and Stafford General Hospital, Staffordshire